CLINICAL TRIAL: NCT06593353
Title: Systems Analysis and Improvement to Optimize Opioid Use Disorder Care Quality and Continuity for Patients Exiting Jail
Acronym: SAIA-MOUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Sarah Odell Gimbel-Sherr, Professor, Child, Family, and Population Health Nursing, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00018542; R01NR021102 (NIH)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder; Opioid Use Disorders
Keywords: Systems Analysis and Improvement Approach (SAIA); Systems Engineering; Medications for Opioid Use Disorder; Continuous Quality Improvement (CQI); Jail; Buprenorphine; implementation science
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: The SAIA (an evidence-based implementation strategy) will be implemented monthly at clinics providing MOUD care. The investigators will apply SAIA at the clinics in Jail Health Services in King County, WA. Those patients who exit jail to the community on MOUD will be tracked to see if they link to any MOUD care services within 30 days. The primary outcome is linkage to MOUD care upon release at any MOUD provider in King County. The secondary outcome assesses whether the patient comes back after initially linking post jail release. SAIA will be implemented in 3 low barrier clinics and the rate of return (sustainment in care -- measured as second visit within 30 days of the first linkage visit will be compared between the three community based MOUD clinics implementing SAIA and all other community-based MOUD clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAIA MOUD clinics in Jail Health Services (Experimental): MOUD clinics within Jail Health Services implementing the Systems Analysis and Improvement Approach (SAIA)
  Interventions: Other: Systems Analysis and Improvement Approach (SAIA)

INTERVENTIONS:
Other: Systems Analysis and Improvement Approach (SAIA) — SAIA an evidence-based, multi-prong, implementation strategy to improve systems thinking amongst frontline care teams to optimize care quality and continuity. The intervention includes monthly meetings where patient care cascades, process mapping and continuous quality improvement are used to identify bottlenecks and prioritize clinic based solutions.

SUMMARY:
This study evaluates the effectiveness of a health systems strategy (the Systems Analysis and Improvement Approach - SAIA) that packages systems engineering tools (including cascade analysis, flow mapping, and continuous quality improvement) to optimize the management of opioid use disorder (MOUD) care cascade and improve linkages between jails and clinical referral sites.

The investigators will

1. study the effectiveness of SAIA on MOUD care cascade quality and continuity for patients receiving care in jail and exiting to referral clinics
2. explore determinants of adoption, implementation, and sustainment of SAIA-MOUD across implementation clinics, and
3. estimate the cost and cost-effectiveness of SAIA-MOUD

DETAILED DESCRIPTION:
SAIA is an evidence-based implementation strategy of bundled systems engineering tools designed to optimize complex healthcare delivery systems and improve linkages between clinical and community providers. The SAIA-MOUD study aims to strengthen the quality and continuity of MOUD care, and linkages to social services, across jail and referral clinics in King County, WA. The investigators will implement the SAIA for three years-including a two-year intensive phase and one year of sustainment-at one jail based MOUD program and three referral MOUD clinics. The investigators will then evaluate the effectiveness of SAIA on improving MOUD cascade quality and continuity for patients receiving care in jail and exiting to referral clinics, determining the effect of SAIA in the jail clinics on linkage to care for community-based MOUD clinics within 30 days of release. A secondary outcome of retention (those who return for a second MOUD pick up within 30 days of initial linkage) will be considered. The investigators will also describe-and explore determinants of-adoption, implementation, and sustainment of SAIA-MOUD via qualitative inquiry with jail and clinic staff. Analysis will be guided by the Consolidated Framework for Implementation Research (CFIR) and the Framework for Reporting Adaptations and Modification to Evidence-based Implementation Strategies (FRAME-IS) will be used to document implementation strategy adaptations. The investigators will estimate the cost and cost-effectiveness of SAIA-MOUD using the cost per quality-adjusted life year gained from the county government, healthcare sector, and societal perspectives. Using a micro-costing approach, the investigators will estimate the incremental costs of implementing and sustaining SAIA in jail and community-based clinics.

ELIGIBILITY:
Inclusion Criteria:

Implementation Outcomes (consented)

Group 1:

* clinic staff/providers at study clinics (JHS, OBOT, Pathways, Sound)
* age 18+

Group 2:

* current patients at SAIA clinic in the community (OBOT, Pathways, Sound) with jail involvement in the last 12 months
* age 18+

Clinical Outcomes (de-identified data, non consented)

Group 3:

* receive MOUD treatment while incarcerated in King County Jails (WA).
* age 18+
* on Medicaid
* released to community

Exclusion Criteria:

Group 1 & 2:

* do not consent

Group 3:

* not on Medicaid

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4165 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Linkage to MOUD Care Upon Release from Jail | 30 days
  the proportion of individuals exiting jails in King County on MOUD who link to any MOUD clinical provider in the community within 30 days

SECONDARY OUTCOMES:
Retention in MOUD Care after Initial Linkage | 30 days
  the proportion of individuals who return for a second MOUD clinical visit within 30 days of initial linkage post jail release

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Odell Gimbel-Sherr, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
The county level data is being sourced from the integrated data hub run by two county level agencies in King County. As a PI, I have requested access but it is not in my rights to give IPD to others, rather it is the right of those who manage the dataset.

REFERENCES:
- [Derived] Gimbel S, Basu A, Callen E, Flaxman AD, Heidari O, Hood JE, Kellogg A, Kern E, Tsui JI, Turley E, Sherr K. Systems analysis and improvement to optimize opioid use disorder care quality and continuity for patients exiting jail (SAIA-MOUD). Implement Sci. 2024 Dec 18;19(1):80. doi: 10.1186/s13012-024-01409-0. PMID 39696305